CLINICAL TRIAL: NCT06311682
Title: A Phase 3 Multi-center Trial to Evaluate the Efficacy and Safety of Tralokinumab in Combination With Topical Corticosteroids in Children (Age 2 to <12 Years) and Infants (Age 6 Months to <2 Years) With Moderate-to-severe Atopic Dermatitis. The Trial is Randomized, Double-blind, Placebo-controlled, and Parallel-group for Children (Age 2 to <12 Years) and Open-label and Single-group for Infants (Age 6 Months to <2 Years)
Brief Title: A Trial to Evaluate the Efficacy and Safety of Tralokinumab in Combination With Topical Corticosteroids in Children and Infants With Moderate-to-severe Atopic Dermatitis
Acronym: TRAPEDS 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LP0162-1336; U1111-1285-6559 (Other: World Health Organization (WHO)); 2023-503630-44-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab; Molasses

STUDY DESIGN:
Intervention Model Description: The study design is parallel for children and a single group for infants.
Who Masked: Participant, Care Provider, Investigator
Masking Description: For subjects aged 2 to <12 years at screening, the trial is double-blind to ensure an objective evaluation of efficacy and safety of the Investigational Medicinal Product (IMP). The subject, the subject's caregiver(s), and the investigator involved in the clinical evaluation and monitoring of the subjects will not be aware of the treatment from baseline to Week 16. However, the site staff that responsible for administering tralokinumab will be aware of the treatment allocation as tralokinumab is visibly different from placebo and has a higher viscosity, requiring more pressure to depress the plunger during injections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tralokinumab + TCS for subjects aged 2 to <12 years (Experimental): Dose and dosing frequency for each subject will depend on the subject's body weight.
  Interventions: Drug: Tralokinumab + TCS
- Placebo + TCS for subjects aged 2 to <12 years (Experimental): Dose and dosing frequency for each subject will depend on the subject's body weight.
  Interventions: Drug: Placebo + TCS
- Tralokinumab + TCS for subjects aged 6 months to <2 years (Experimental): Dose and dosing frequency for each subject will depend on the subject's body weight.
  Interventions: Drug: Tralokinumab + TCS

INTERVENTIONS:
Drug: Tralokinumab + TCS — The trial medication will be given under the skin (SC). Dose and dosing frequency for each subject will depend on the subject's body weight. Subjects who will receive treatment every two weeks will receive a loading dose corresponding to a double dose at baseline. Subjects who will receive treatment every 4 weeks will receive a staggered loading dose at baseline and Week 2. After the loading dose, they will continue to receive treatment every 4 weeks. The dose and dosing frequency will be adjusted according to the subject's body weight at weeks 16, 32, 52, 64, 88, 112, 136, 160, and 184.
  Arms: Tralokinumab + TCS for subjects aged 2 to <12 years; Tralokinumab + TCS for subjects aged 6 months to <2 years
Drug: Placebo + TCS — The trial medication will be given under the skin (SC). Dose and dosing frequency for each subject will depend on the subject's body weight. Subjects who will receive treatment every two weeks will receive a loading dose corresponding to a double dose at baseline. Subjects who will receive treatment every 4 weeks will receive a staggered loading dose at baseline and Week 2. After the loading dose, they will continue to receive treatment every 4 weeks. The dose and dosing frequency will be adjusted according to the subject's body weight at weeks 16, 32, 52, 64, 88, 112, 136, 160, and 184.
  Arms: Placebo + TCS for subjects aged 2 to <12 years

SUMMARY:
The purpose of this trial is to test whether treatment with tralokinumab (administered subcutaneous injections [SC]) in combination with topical corticosteroids (TCS) is safe and effective to treat moderate-to-severe atopic dermatitis (AD) in children and infants. This will be judged by a range of assessments that rate the severity and extent of atopic dermatitis and its symptoms, as well as general health status and quality of life. The trial will last for up to 4 years. There will be visits every 2 weeks for the first year and every 6 weeks thereafter. Some of the visits will be conducted by phone.

The study involves two different age groups: children aged 2 to under 12 years and infants aged 6 months to under 2 years. This trial compares tralokinumab +TCS to placebo + TCS for children with moderate-to-severe AD and evaluates tralokinumab + TCS for infants with moderate-to-severe AD. Infants will not receive placebo. All subjects will go through a screening process, which is the first part of the trial and will last up to 4 weeks. During this period, it will be checked if the child or infant meets the criteria to participate in the trial.

The children will be randomly assigned to receive tralokinumab + TCS or placebo + TCS for the initial 16 weeks, with the treatment being double-blinded. During the first 16 weeks, children will have a 2 out of 3 chance of getting tralokinumab and a 1 out of 3 chance of getting placebo. Thereafter, all subjects will receive tralokinumab + TCS. The infants will receive tralokinumab + TCS as open-label treatment for the entire treatment period, meaning that the participants will know they are receiving tralokinumab. After stopping treatment, all participants will enter a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to <12 years at screening.
* Body weight ≥9 kg at screening.
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD.
* History of AD for: ≥12 months for subjects aged ≥6 years at screening and ≥3 months for subjects aged 6 months to <6 years at screening.
* Documented inadequate response to mid-strength TCS within 6 months before the screening visit.
* AD involvement of ≥10% body surface area at screening and baseline according to component A of SCORAD.
* An EASI score of ≥16 at screening and baseline.
* An IGA score of ≥3 at screening and baseline.
* A Child Worst Itch NRS average score of ≥4 (subjects aged ≥6 years at screening) or a Scratch ObsRO average score of ≥4 (subjects aged <6 years at screening) during the week prior to baseline.

Exclusion Criteria:

* Treatment with the topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), topical phosphodiesterase-4 inhibitors (PDE-4), and topical Janus kinase inhibitors (JAK) within 1 week prior to baseline.
* Treatment with bleach baths within 1 week prior to baseline.
* Treatment with the immunomodulatory medications systemic immunosuppressive/immunomodulating drugs (e.g. methotrexate, cyclosporine, azathioprine, mycophenolate mofetil, Janus kinase inhibitors) and systemic corticosteroids (excludes inhaled, ophthalmic, or intranasal delivery) within 4 weeks prior to baseline.
* Use of tanning beds or phototherapy within 4 weeks prior to baseline.
* Treatment with a live (attenuated) or non-live vaccine within 30 days prior to the baseline visit.
* Active dermatologic conditions that may confound the diagnosis of AD or would interfere with assessment of treatment such as seborrheic dermatitis, active skin infection, scabies, cutaneous T cell lymphoma, or psoriasis.
* Clinically significant active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antifungals or antiprotozoal within 2 weeks before the baseline visit.
* History of past or current hepatitis B or C including a positive hepatitis B or C test at screening.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 2 to <12 years at screening. | At week 16
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.

SECONDARY OUTCOMES:
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 6 month to <2 years at screening. | At week 16
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 50% reduction in EASI score in subjects aged 2 to <12 years at screening. | At week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 50% reduction in EASI score in subjects aged 6 month to <2 years at screening. | At week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 2 to <12 years at screening. | From baseline to week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in Scoring Atopic Dermatitis (SCORAD) in subjects aged 2 to <12 years at screening. | From baseline to week 16
  The SCORAD is a validated tool to evaluate the extent and severity of atopic dermatitis. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  The SCORAD is a validated tool to evaluate the extent and severity of atopic dermatitis. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in affected BSA in subjects aged 2 to <12 years at screening. | From baseline to week 16
  BSA is a body surface area.
Percent change in affected BSA in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  BSA is a body surface area.
Percent change in Children's Dermatology Life Quality Index (CDLQI) for subjects aged 4 to <12 years at screening. | From baseline to Week 16
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Reduction in Child Worst Itch numeric rating score (NRS) (weekly average) ≥4 for subjects aged 6 to <12 years at screening. | From baseline to Week 16
  The Child Worst Itch NRS assesses 'worst itch today' and 'worst itch last night' using a numerical rating scale from 0 to 10, where 0 represents 'Not itchy at all' and 10 represents 'Very itchy'.
Reduction in Scratch Observer-Reported Outcome (ObsRO) (weekly average) ≥4 for subjects aged 2 to <6 years at screening. | From baseline to week 16
  The Scratch ObsRO NRS assesses 'worst scratching during the past 24 hours' using a numerical rating scale from 0 to 10, where 0 represents 'No scratching' and 10 represents 'Worst scratching possible'.
Reduction in Scratch Observer-Reported Outcome (ObsRO) (weekly average) ≥4 for subjects aged 6 months to <2 years years at screening. | From baseline to week 16
  The Scratch ObsRO NRS assesses 'worst scratching during the past 24 hours' using a numerical rating scale from 0 to 10, where 0 represents 'No scratching' and 10 represents 'Worst scratching possible'.
Reduction of ≥4 in Child Worst Itch NRS (weekly average) for subjects aged 6 to <12 years at screening or Scratch ObsRO (weekly average) for subjects aged 2 to <6 years at screening. | From baseline to week 16
  The Child Worst Itch NRS assesses 'worst itch today' and 'worst itch last night' using a numerical rating scale from 0 to 10, where 0 represents 'Not itchy at all' and 10 represents 'Very itchy'.
  The Scratch ObsRO NRS assesses 'worst scratching during the past 24 hours' using a numerical rating scale from 0 to 10, where 0 represents 'No scratching' and 10 represents 'Worst scratching possible'.
Percent change in Patient-Oriented Eczema Measure (POEM) in subjects aged 2 to <12 years at screening. | From baseline to week 16
  The POEM is a validated questionnaire used to assess disease symptoms in atopic eczema patients in both clinical practice and clinical trials. The tool consists of 7 items each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Subjects will score how often they have experienced each symptom over the previous week on a 5-point categorical response scale (0 = 'no days'; 1 = '1 to 2 days'; 2 = '3 to 4 days'; 3 = '5 to 6'days; 4 = 'every day'). The total score is the sum of the 7 items (range 0 to 28) and reflects disease-related morbidity; a high score is indicative of a worse disease severity.
Percent change in Patient-Oriented Eczema Measure (POEM) in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  The POEM is a validated questionnaire used to assess disease symptoms in atopic eczema patients in both clinical practice and clinical trials. The tool consists of 7 items each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Subjects will score how often they have experienced each symptom over the previous week on a 5-point categorical response scale (0 = 'no days'; 1 = '1 to 2 days'; 2 = '3 to 4 days'; 3 = '5 to 6'days; 4 = 'every day'). The total score is the sum of the 7 items (range 0 to 28) and reflects disease-related morbidity; a high score is indicative of a worse disease severity.
Reduction of in Patient-Oriented Eczema Measure (POEM) ≥6 in subjects aged 2 to <12 years at screening. | From baseline to week 16
  The POEM is a validated questionnaire used to assess disease symptoms in atopic eczema patients in both clinical practice and clinical trials. The tool consists of 7 items each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Subjects will score how often they have experienced each symptom over the previous week on a 5-point categorical response scale (0 = 'no days'; 1 = '1 to 2 days'; 2 = '3 to 4 days'; 3 = '5 to 6'days; 4 = 'every day'). The total score is the sum of the 7 items (range 0 to 28) and reflects disease-related morbidity; a high score is indicative of a worse disease severity.
Reduction of in Patient-Oriented Eczema Measure (POEM) ≥6 in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  The POEM is a validated questionnaire used to assess disease symptoms in atopic eczema patients in both clinical practice and clinical trials. The tool consists of 7 items each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Subjects will score how often they have experienced each symptom over the previous week on a 5-point categorical response scale (0 = 'no days'; 1 = '1 to 2 days'; 2 = '3 to 4 days'; 3 = '5 to 6'days; 4 = 'every day'). The total score is the sum of the 7 items (range 0 to 28) and reflects disease-related morbidity; a high score is indicative of a worse disease severity.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 2 to <12 years at screening. | From baseline to week 16
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Change in Child Worst Itch NRS (weekly average) for subjects aged 6 to <12 years at screening. | From baseline to week 16
  The Scratch ObsRO NRS assesses 'worst scratching during the past 24 hours' using a numerical rating scale from 0 to 10, where 0 represents 'No scratching' and 10 represents 'Worst scratching possible'.
Change in Scratch Observer-Reported Outcome (ObsRO) (weekly average) in subjects aged 2 to <6 years at screening. | From baseline to week 16
  The Scratch ObsRO NRS assesses 'worst scratching during the past 24 hours' using a numerical rating scale from 0 to 10, where 0 represents 'No scratching' and 10 represents 'Worst scratching possible'.
Change in Scratch Observer-Reported Outcome (ObsRO) (weekly average) in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  The Scratch ObsRO NRS assesses 'worst scratching during the past 24 hours' using a numerical rating scale from 0 to 10, where 0 represents 'No scratching' and 10 represents 'Worst scratching possible'.
Reduction in Children's Dermatology Life Quality Index (CDLQI) ≥6 for subjects aged 4 to <12 years at screening. | From baseline to week 16
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Number of treatment-emergent adverse events (AEs) per subject aged 2 to <12 years at screening. | From baseline to week 16
  An adverse event (AE) is any unexpected medical issue that happens to a person who is taking a medication or participating in a study. It could be a symptom, disease, or abnormal test result, even if it's not necessarily caused by the medication being used.
Number of treatment-emergent adverse events (AEs) per subject aged 6 month to <2 years at screening. | From baseline to week 16
  An adverse event (AE) is any unexpected medical issue that happens to a person who is taking a medication or participating in a study. It could be a symptom, disease, or abnormal test result, even if it's not necessarily caused by the medication being used.
Presence of treatment-emergent anti-drug antibodies (yes/no) in subjects aged 2 to <12 years at screening. | From baseline to week 16
Presence of treatment-emergent anti-drug antibodies (yes/no) in subjects aged 6 month to <2 years at screening. | From baseline to week 16
Rescue treatment use (yes/no) in subjects aged 2 to <12 years at screening. | From baseline to week 16
Rescue treatment use (yes/no) in subjects aged 6 month to <2 years at screening. | From baseline to week 16
Number of TCS free days in subjects aged 2 to <12 years at screening. | From baseline to week 16
  TCS- tropical corticosteroids.
Number of TCS free days in subjects aged 6 month to <2 years at screening. | From baseline to week 16
  TCS- tropical corticosteroids.
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 2 to <12 years at screening. | At week 52
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 6 month to <2 years at screening. | At week 52
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 52
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 52
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 52
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 52
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 2 to <12 years at screening. | From baseline to week 52
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 6 month to <2 years at screening. | From baseline to week 52
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in Scoring Atopic Dermatitis (SCORAD) in subjects aged 2 to <12 years at screening. | From baseline to week 52
  The SCORAD is a validated tool to evaluate the extent and severity of atopic dermatitis. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) in subjects aged 6 month to <2 years at screening. | From baseline to week 52
  The SCORAD is a validated tool to evaluate the extent and severity of atopic dermatitis. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in affected body surface area (BSA) in subjects aged 2 to <12 years at screening. | From baseline to week 52
Percent change in affected body surface area (BSA) in subjects aged 6 month to <2 years at screening. | From baseline to week 52
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 2 to <12 years at screening. | From baseline to week 52
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 6 month to <2 years at screening. | From baseline to week 52
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Children's Dermatology Life Quality Index (CDLQI) in subjects aged 4 to <12 years at screening. | From baseline to week 52
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Reduction in Children's Dermatology Life Quality Index (CDLQI) ≥6 for subjects aged 4 to <12 years at screening. | From baseline to week 52
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Reduction of in Patient-Oriented Eczema Measure (POEM) ≥6 in subjects aged 2 to <12 years at screening. | From baseline to week 52
  The POEM is a validated questionnaire used to assess disease symptoms in atopic eczema patients in both clinical practice and clinical trials. The tool consists of 7 items each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Subjects will score how often they have experienced each symptom over the previous week on a 5-point categorical response scale (0 = 'no days'; 1 = '1 to 2 days'; 2 = '3 to 4 days'; 3 = '5 to 6'days; 4 = 'every day'). The total score is the sum of the 7 items (range 0 to 28) and reflects disease-related morbidity; a high score is indicative of a worse disease severity.
Reduction of in Patient-Oriented Eczema Measure (POEM) ≥6 in subjects aged 6 month to <2 years at screening. | From baseline to week 52
  The POEM is a validated questionnaire used to assess disease symptoms in atopic eczema patients in both clinical practice and clinical trials. The tool consists of 7 items each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Subjects will score how often they have experienced each symptom over the previous week on a 5-point categorical response scale (0 = 'no days'; 1 = '1 to 2 days'; 2 = '3 to 4 days'; 3 = '5 to 6'days; 4 = 'every day'). The total score is the sum of the 7 items (range 0 to 28) and reflects disease-related morbidity; a high score is indicative of a worse disease severity.
Number of treatment-emergent adverse events (AEs) per subject aged 2 to <12 years at screening. | From week 16 to 52
  An adverse event (AE) is any unexpected medical issue that happens to a person who is taking a medication or participating in a study. It could be a symptom, disease, or abnormal test result, even if it's not necessarily caused by the medication being used.
Number of treatment-emergent adverse events (AEs) per subject aged 6 month to <2 years at screening. | From week 16 to 52
  An adverse event (AE) is any unexpected medical issue that happens to a person who is taking a medication or participating in a study. It could be a symptom, disease, or abnormal test result, even if it's not necessarily caused by the medication being used.
Presence of treatment-emergent anti-drug antibodies (yes/no) in subjects aged 2 to <12 years at screening. | From week 16 to 52
  It measures whether the developed antibodies in response to the treatment have any effect on the safety and effectiveness of the treatment.
Presence of treatment-emergent anti-drug antibodies (yes/no) in subjects aged 6 month to <2 years at screening. | From week 16 to 52
  It measures whether the developed antibodies in response to the treatment have any effect on the safety and effectiveness of the treatment.
Number of treatment-emergent adverse events (AEs) per subject aged 2 to <12 years at screening. | From week 52 to end of treatment
  An adverse event (AE) is any unexpected medical issue that happens to a person who is taking a medication or participating in a study. It could be a symptom, disease, or abnormal test result, even if it's not necessarily caused by the medication being used.
Number of treatment-emergent adverse events (AEs) per subject aged 6 month to <2 years at screening. | From week 52 to end of treatment
  An adverse event (AE) is any unexpected medical issue that happens to a person who is taking a medication or participating in a study. It could be a symptom, disease, or abnormal test result, even if it's not necessarily caused by the medication being used.
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 2 to <12 years at screening. | At week 100
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 6 month to <2 years at screening. | At week 100
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 100
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 100
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 100
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 100
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 2 to <12 years at screening. | From baseline to week 100
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 6 month to <2 years at screening. | From baseline to week 100
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 2 to <12 years at screening. | From baseline to week 100
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 6 month to <2 years at screening. | From baseline to week 100
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Children's Dermatology Life Quality Index (CDLQI) for subjects aged 4 to <12 years at screening. | From baseline to week 100
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Reduction in Children's Dermatology Life Quality Index (CDLQI) ≥ 6 for subjects aged 4 to <12 years at screening. | From baseline to week 100
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 2 to <12 years at screening. | At week 148
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 6 month to <2 years at screening. | At week 148
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 148
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 148
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 148
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 148
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 2 to <12 years at screening. | From baseline to week 148
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 6 month to <2 years at screening. | From baseline to week 148
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 2 to <12 years at screening. | From baseline to week 148
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 6 month to <2 years at screening. | From baseline to week 148
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Children's Dermatology Life Quality Index (CDLQI) for subjects aged 4 to <12 years at screening. | From baseline to week 148
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Reduction in Children's Dermatology Life Quality Index (CDLQI) ≥ 6 for subjects aged 4 to <12 years at screening. | From baseline to week 148
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 2 to <12 years at screening. | At week 196
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Investigator's Global Assessment for atopic dermatitis (IGA 0/1) score of 0 (clear) or 1 (almost clear) in subjects aged 6 month to <2 years at screening. | At week 196
  The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 196
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 75% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 196
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 2 to <12 years at screening. | At week 196
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Having at least 90% reduction in Eczema Area and Severity Index (EASI) score in subjects aged 6 month to <2 years at screening. | At week 196
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 2 to <12 years at screening. | From baseline to week 196
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in EASI in subjects aged 6 month to <2 years at screening. | From baseline to week 196
  The EASI is a validated measure to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 2 to <12 years at screening. | From baseline to week 196
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) sleep loss in subjects aged 6 month to <2 years at screening. | From baseline to week 196
  The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Percent change in Children's Dermatology Life Quality Index (CDLQI) for subjects aged 4 to <12 years at screening. | From baseline to week 196
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Reduction in Children's Dermatology Life Quality Index (CDLQI) ≥ 6 for subjects aged 4 to <12 years at screening. | From baseline to week 196
  The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (61):
- United States (14):
  - Leo Pharma Investigational site, Birmingham, Alabama
  - Leo Pharma Investigational site, North Little Rock, Arkansas
  - Leo Pharma Investigational site, Palo Alto, California
  - Leo Pharma Investigational site, Sacramento, California
  - Leo Pharma Investigational site, San Diego, California
  - Leo Pharma Investigational site, Jacksonville, Florida
  - Leo Pharma Investigational site, Miami, Florida
  - Leo Pharma Investigational site, Tampa, Florida
  - Leo Pharma Investigational site, Macon, Georgia
  - Leo Pharma Investigational site, Waterford, Michigan
  - Leo Pharma Investigational site, Tulsa, Oklahoma
  - Leo Pharma Investigational site, Portland, Oregon
  - Leo Pharma Investigational site, Charleston, South Carolina
  - Leo Pharma Investigational site, Norfolk, Virginia
- Belgium (4):
  - Leo Pharma Investigational site, Brussels
  - Leo Pharma Investigational site, Ghent
  - Leo Pharma Investigational site, Leuven
  - Leo Pharma Investigational site, Liège
- Canada (8):
  - Leo Pharma Investigational site, Burlington
  - Leo Pharma Investigational site, Calgary
  - Leo Pharma Investigational site, Edmonton
  - Leo Pharma Investigational site, Hamilton
  - Leo Pharma Investigational site, Niagara Falls
  - Leo Pharma Investigational site, Saskatoon
  - Leo Pharma Investigational site, Windsor
  - Leo Pharma Investigational site, Winnipeg
- Croatia (2):
  - Leo Pharma Investigational site, Rijeka
  - Leo Pharma Investigational site, Zagreb
- Germany (6):
  - Leo Pharma Investigational site, Buxtehude
  - Leo Pharma Investigational site, Dresden
  - Leo Pharma Investigational site, Mainz
  - Leo Pharma Investigational site, Osnabrück
  - Leo Pharma Investigational site, Tübingen
  - Leo Pharma Investigational site, Wuppertal
- Ireland (2):
  - Leo Pharma Investigational site, Cork
  - Leo Pharma Investigational site, Crumlin
- Italy (5):
  - Leo Pharma Investigational site, Ancona
  - Leo Pharma Investigational site, Brescia
  - Leo Pharma Investigational site, Padua
  - Leo Pharma Investigational site, Roma
  - Leo Pharma Investigational site, Rome
- Leo Pharma Investigational site, Utrecht, Netherlands
- Poland (7):
  - Leo Pharma Investigational site, Gdansk
  - Leo Pharma Investigational site, Krakow
  - Leo Pharma Investigational site, Lodz
  - Leo Pharma Investigational site, Ostrowiec Świętokrzyski
  - Leo Pharma Investigational site, Rzeszów
  - Leo Pharma Investigational site, Tarnów
  - Leo Pharma Investigational site, Warsaw
- Romania (2):
  - Leo Pharma Investigational site, Brasov
  - Leo Pharma Investigational site, Iași
- South Korea (3):
  - Leo Pharma Investigational site, Ansan-si
  - Leo Pharma Investigational site, Gwangju
  - Leo Pharma Investigational site, Seoul
- Spain (3):
  - Leo Pharma Investigational site, Alicante
  - Leo Pharma Investigational site, Madrid
  - Leo Pharma Investigational site, Valencia
- United Kingdom (4):
  - Leo Pharma Investigational site, Lincoln
  - Leo Pharma Investigational site, London
  - Leo Pharma Investigational site, Sheffield
  - Leo Pharma Investigational site, Southampton

IPD SHARING:
Plan to Share IPD: No